CLINICAL TRIAL: NCT00378274
Title: Pain, Anxiety and Depression in Chronic Pain Patients With and Without Neuropathic Pain Compared With Healthy Volunteers
Brief Title: Descriptive Study of Pain, Anxiety and Depression
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Other Study IDs: KVA2006LG
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2007-11-16 (Estimated); Status verified 2007-11

CONDITIONS: Pain
Keywords: Neuropathic pain; Chronic pain; Depression; Anxiety
MeSH Terms: conditions — Pain; Neuralgia; Chronic Pain; Depression; Anxiety Disorders | interventions — Observation

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Observation

SUMMARY:
The purpose of the study is to investigate pain, anxiety and depression in chronic pain patients with and without neuropathic pain compared with healthy volunteers

DETAILED DESCRIPTION:
Primary outcome measures:

* Symptom checklist 92

Secondary outcome measures:

* Hamilton Depression and Anxiety Rating Scale
* Major Depression Inventory
* GAD-10 Anxiety Scale
* Health Survey SF-36
* McGill Pain Questionnaire
* Sweat test
* Heart rate variability testing
* Coping Strategy Questionnare
* Quantitative sensory testing
* Pain Catastrophizing Scale
* Pain rating (VAS)
* Interview

ELIGIBILITY:
Inclusion Criteria:

* Neuropathic pain patient or patient with fibromyalgia
* Daily pain in more than 6 months
* Weekly average pain score 4 or more (VAS)

Exclusion Criteria:

* Treatment with antidepressants, anticonvulsants or any other pain medication except paracetamol
* Serious or unstable medical disease
* Prior or present diagnosis of mania, bipolar or psychotic disorder, delirium, suicidal, drug and alcohol dependence, severe agitation
* Patients who cannot cooperate and do not understand Danish

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-09; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Gormsen, MD, Principal Investigator — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark